CLINICAL TRIAL: NCT01612390
Title: Comparison of Sublingual Misoprostol and Intravenous Oxytocin in Active Management of the Third Stage of Labor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rasha Mohammed Mohammed Badawi (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Rasha Mohammed Mohammed Badawi, RBadawi, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: hit 1234
Record Dates: First submitted 2012-06-02; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Postpartum Hemorrhage Prevention by Using Oxytocin Verses Misoprostol
Keywords: postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- group 1: receive 400 Mg sublingual misoprostol.
- group 2: receive 600 Mg sublingual misoprostol.
- group 3: receive 5IU of intravenous oxytocin.

SUMMARY:
Sublingual misoprostol is superior to oxytocin in reduction of blood loss during the third and fourth stages of labor

DETAILED DESCRIPTION:
Sublingual misoprostol is superior to oxytocin in reduction of blood loss during the third and fourth stages of labor as The data from a pharmacokinetics study suggested that the bioavaiblitiy of misoprostol after sub-lingual administration was higher than those after oral or vaginal administration

ELIGIBILITY:
Inclusion Criteria:

* Women with aheathy singleton pregnancy in spontaneous or induced labor at term .

Exclusion Criteria:

* Hypersensitivity/Contraindication to prostaglandins Antepartum hemorrhage Multiple pregnancy Cardiac disease Malpresentation Rhesus- negative mother hypersensitive disorders Severe anaemia(hemoglobin<7g/dl)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include (180)randomly allocated
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
reduce blood loss during third and fourth stages of labor. | 1 year
  reduce blood loss during third and fourth stages of labor by using misopristol is better than using oxytocin

SECONDARY OUTCOMES:
the duration of the third stage of labor ,need for oxytocics ,blood transfusion and any adverse effects of the drugs | 1 year
  the duration of the third stage of labor ,needed for oxytocics ,blood transfusion and any adverse effects of the drug will be reduced with mesopristol

CONTACTS AND LOCATIONS:
Overall Officials: RBadawi mohamed, M.B;B.CH, Principal Investigator — Ain Shams University
Locations (1):
- AinShamsU, Cairo, Egypt